CLINICAL TRIAL: NCT05455502
Title: A Phase 1, Open-label, Randomized, Crossover Study to Evaluate the Relative Bioavailability and Food Effect of a New Tablet Formulation of VX-548 in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Relative Bioavailability and Food Effect of a New Tablet Formulation of VX-548
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VX21-548-011
Record Dates: First submitted 2022-07-07; First posted 2022-07-13 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Participants will receive VX-548 reference tablet (TF1) under fasted condition in dosing period 1, then VX-548 test tablet (TF2) under fasted condition in dosing period 2, and finally VX-548 test tablet (TF2) under fed condition in dosing period 3. A washout period of 12 days will be maintained between 3 dosing periods.
  Interventions: Drug: VX-548
- Sequence 2 (Experimental): Participants will receive VX-548 TF1 under fasted condition in dosing period 1, then VX-548 TF2 under fed condition in dosing period 2, and finally VX-548 TF2 under fasted condition in dosing period 3. A washout period of 12 days will be maintained between 3 dosing periods.
  Interventions: Drug: VX-548
- Sequence 3 (Experimental): Participants will receive VX-548 TF2 under fasted condition in dosing period 1, then VX-548 TF1 under fasted condition in dosing period 2, and finally VX-548 TF2 under fed condition in dosing period 3. A washout period of 12 days will be maintained between 3 dosing periods.
  Interventions: Drug: VX-548
- Sequence 4 (Experimental): Participants will receive VX-548 TF2 under fasted condition in dosing period 1, then VX-548 TF2 under fed condition in dosing period 2, and finally VX-548 TF1 under fasted condition in dosing period 3. A washout period of 12 days will be maintained between 3 dosing periods.
  Interventions: Drug: VX-548
- Sequence 5 (Experimental): Participants will receive VX-548 TF2 under fed condition in dosing period 1, then VX-548 TF1 under fasted condition in dosing period 2, and finally VX-548 TF2 under fasted condition in dosing period 3. A washout period of 12 days will be maintained between 3 dosing periods.
  Interventions: Drug: VX-548
- Sequence 6 (Experimental): Participants will receive VX-548 TF2 under fed condition in dosing period 1, then VX-548 TF2 under fasted condition in dosing period 2, and finally VX-548 TF1 under fasted condition in dosing period 3. A washout period of 12 days will be maintained between 3 dosing periods.
  Interventions: Drug: VX-548

INTERVENTIONS:
Drug: VX-548 — Tablet for oral administration.
  Other Names: Suzetrigine

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability and food effect of a new tablet formulation of VX-548 in healthy adult participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4) (A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (Kg/m^2)
* A total body weight greater than (>)50 kg

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption
* Female participants of childbearing potential
* Male participants with a female partner who is pregnant, nursing, or planning to become pregnant during the study
* History of cardiovascular disease, cardiac dysrhythmias or central nervous system disease

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2022-09-17 (Actual); Study Completion 2022-09-17 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of VX-548 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 144, up to 216 hours Post-dose
Area Under the Concentration Versus Time Curve From the Time of Dosing to the Last Measurable Concentration (AUClast) of VX-548 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 144, up to 216 hours Post-dose
Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of VX-548 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 144, up to 216 hours Post-dose

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of VX-548 Metabolite | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 144, up to 216 hours Post-dose
Area Under the Concentration Versus Time Curve From the Time of Dosing to the Last Measurable Concentration (AUClast) of VX-548 Metabolite | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 144, up to 216 hours Post-dose
Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of VX-548 Metabolite | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 144, up to 216 hours Post-dose
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Day 40

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Salt Lake City, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing